# Cover Page

Title of the Study: Consumer Motivation for Disease Prevention

NCT number: Not available

Date of Document: April 2, 2019.

Document Type: Statistical Analysis Plan

## Methodology:

Randomized Lab Study. All responses are to be collected within a single survey session.

## Sampling Frame:

Student sample (university students who participate in the study in exchange for course credits)

Design: The study has a 2 (presence of uncontrollable factor: yes vs. no)  $\times$  2 (Anticipated regret induction: yes vs. no) between-subject design. Participants will be randomly assigned to one of the 4 between-subject conditions.

There is also a within-subject variable. Each subject will respond to 10 rounds of decision task with 5 different levels of overall disease risk reduction brought by the removal of X. The 5 levels of risk reduction are: (i) Removal of X reduces disease risk from 60% to 50%; (ii) 60% to 40%; (iii) 60% to 20%; (v) 60% to 10%.

#### Randomization:

Participants will be randomly assigned to one of the 4 between-subject arms. Randomization will be performed using the built-in algorithm in Z-tree (computer software).

#### Attrition:

No attrition expected. Because the study will involve only one 30-minute survey session, all participants are expected to finish the survey.

## Statistical Analysis plan:

Primary Outcome (Decision to remove X): Logistic regression will be conducted using the decision to remove X(1/0) as the dependent variable and the three variables — presence of uncontrollable risk factor, anticipated regret induction, and magnitude of overall risk reduction — as the independent variables.

## **Secondary Outcomes:**

ANOVA will be conducted for each of the three psychological measures. Independent variables are presence of uncontrollable risk factor and anticipated regret induction.